CLINICAL TRIAL: NCT06375811
Title: Pre-IVF Treatment With a GnRH Antagonist in Women With Endometriosis - A Prospective Clinical Trial
Brief Title: Pre-IVF Treatment With a GnRH Antagonist in Women With endometriosis_temp
Acronym: PREGnant
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: University of Colorado, Denver (Other); Northwestern University (Other); University of North Carolina (Other); Duke University (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Heping Zhang, professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2000027121_a
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Infertility; Endometriosis
MeSH Terms: conditions — Infertility; Endometriosis | interventions — elagolix

STUDY DESIGN:
Intervention Model Description: Half of the subjects (200, randomized or not randomized) will receive elagolix 200mg twice a day (BID) and the other half of subjects will receive placebo BID or SOC IVF (200, placebo or SOC IVF). Elagolix or placebo will be taken for a minimum of 60 days before IVF cycle start. For convenience of IVF cycle scheduling, participants may receive up to an additional 14 days of intervention (elagolix or placebo) beyond the minimum 60 days of pre-IVF treatment, such that the last dose of study intervention (elagolix or placebo) is received no more than 24 hours before start of IVF treatment protocol.
Who Masked: Participant, Care Provider, Investigator
Masking Description: For participants who agree to be randomized, a computer-generated randomization list will be created by the PREGnant Data Coordinating Center (DCC) and randomization will be performed prior to the first dose of elagolix. Randomization will have random sizes (2, 4, or 6) of blocks and be stratified by site, i.e. whole blocks are assigned to sites. The randomization list will not be available to any person involved in the conduct and evaluation of the trial until the trial is complete and database is declared clean and is released by the DCC. Likewise, treatment allocation information will not be accessible to investigators (except for serious safety concerns), trial staff at the site or central laboratory personnel during the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-IVF Treatment with 60 day course of oral GnRH antagonist (Active Comparator): For those who agree to be randomized, subjects will be randomized to elagolix 200mg BID. The medication will be taken orally and subjects will be counseled to take the medication at the same time each day. This arm will also include participants who do not want to be randomized while choose elagolix.
  Interventions: Drug: Elagolix 200 MG
- Pre-IVF Treatment with 60 day course of Placebo or SOC IVF (Other): For those who agree to be randomized, subjects will be randomized to placebo, BID. The medication will be taken orally and subjects will be counseled to take the medication at the same time each day. This arm will also include participants who want to continue their ongoing or planned IVF and follow standard of care (SOC) (SOC IVF) if the participants do not want to delay the IVF procedure.
  Interventions: Other: Placebo or SOC IVF

INTERVENTIONS:
Drug: Elagolix 200 MG — Elagolix tablet
  Other Names: Orlissa
  Arms: Pre-IVF Treatment with 60 day course of oral GnRH antagonist
Other: Placebo or SOC IVF — Sugar pill manufactured to mimic Elagolix 200mg
  Arms: Pre-IVF Treatment with 60 day course of Placebo or SOC IVF

SUMMARY:
A Phase 3 clinical trial of oral GnRH antagonist pre-treatment for women with endometriosis who are undergoing IVF, with a primary outcome of live birth rate. The investigators' central hypothesis is that in infertile woman with endometriosis undergoing in vitro fertilization-embryo transfer (IVF-ET), live birth rates will improve in those pretreated with GnRH antagonist compared to those not pretreated with GnRH antagonist.

DETAILED DESCRIPTION:
Infertility is a common complication of endometriosis; while IVF successfully treats endometriosis-associated infertility, pregnancy rates are diminished compared to other etiologies of infertility. The study's long- term objectives are to better identify and treat endometriosis related infertility. The investigators' central hypothesis is that in infertile woman with endometriosis undergoing in vitro fertilization-embryo transfer (IVF-ET), live birth rates will improve in those pretreated with GnRH antagonist compared to those not pretreated with GnRH antagonist. The use of gonadotropin releasing hormone (GnRH) agonist prior to IVF has been suggested to improve success, however studies have been small and rarely reported live birth rates. Further, use of this approach is limited by the long treatment time required. Recent approval of an oral GnRH antagonist for endometriosis provides a novel option for women with endometriosis who are undergoing IVF. This agent avoids parenteral administration and the prolonged delay in initiation of action as was seen with GnRH agonists. There have been no studies on the efficacy of GnRH antagonists for the treatment of endometriosis-related infertility. The investigators propose a clinical trial of oral GnRH antagonist pre-treatment for women with endometriosis who are undergoing IVF, with a primary outcome of live birth rate. Participants will include those who agree to be randomized and those who do not want to be randomized. Those who agree to be randomized will be randomly assigned to either the elagolix group or placebo group. Those who do not want to be randomized can choose either the active treatment elagolix and follow the same procedures as those agreeing to be randomized or continue their ongoing or planned IVF and follow standard of care (SOC) (SOC IVF) if they do not want to delay the IVF procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Women who plan to undergo IVF for treatment of infertility.
2. Age ≥18 and <40 years at time of egg retrieval or signing informed consent.
3. Documentation of diagnosis of endometriosis by surgical visualization of endometriosis (laparoscopy or laparotomy) or diagnosis by pathology within the last 10 years before the initial trial entry visit or documentation of ovarian endometrioma >2 cm or two or more smaller endometriomas that total >2 cm in diameter. If entry is based on the presence of an endometrioma, transvaginal ultrasound evaluation must document the same unambiguous endometrioma on two separate occasions in more than one menstrual cycle. Images will be printed or transmitted electronically and read centrally by investigators at Yale to assure uniform diagnostic criteria (classic ground glass appearance) are applied.
4. Body mass index (BMI) of 18-40 kg/m2 (both inclusive) at screening.
5. AMH > 0.5ng/ml, within 12 months of a fresh IVF cycle start. For frozen embryo transfers (FET) , AMH level eligibility criteria may not be met as long as the patient has at least one good quality blastocyst stored for the FET.
6. No known uterine cavity abnormalities at time of screening. Uterine cavity assessment by sonohysterogram or hysteroscopy within 12 months of embryo transfer indicating absence of focal intracavitary pathology and hence establishing adequate cavity at the time of embryo transfer. Ultrasound or MRI features suggestive of adenomyosis will be acceptable for inclusion. Type 3 fibroids are allowed up to 4cm size.
7. Presence of at least one ovary with no clinically significant abnormalities other than endometrioma. For eligible women with evidence of a hemorrhagic ovarian cyst, a repeat US will be needed in a subsequent menstrual cycle to ensure persistent cyst for patient to be deemed eligible.
8. Negative urine or cervical swab for gonorrhea and chlamydia within 12 months of screening.
9. Willing and able to comply with trial procedures, including reporting of obstetrical outcomes after delivery.

Exclusion Criteria:

1. Use of depot GnRH agonists within 6 months of study start. Use of subcutaneous antagonists or nasal agonist within 2 months of study start unless part of regular IVF or previous IUI cycle°.
2. Use of depot medroxyprogesterone acetate (MPA) (injectable) or birth control implants (e.g., Implanon® or Nexplanon®) within 6 months of study start°.
3. Continuous use of oral progestins (MPA, NETA) within 1 month of study start°.
4. Use of aromatase inhibitors, danazol or hormonal contraceptives (Including combined oral contraceptive pill, progestin-only pill, transdermal patch or contraceptive ring, or double barrier contraception) within 1 month of study start.
5. Pregnancy greater than 8 weeks in length within the last 6 months.
6. Number of previous IVF/ICSI attempts ≥3 unsuccessful (negative pregnancy test).
7. Presence of hydrosalpinx measuring >2cm on ultrasound, untreated endometrial polyps or intrauterine adhesions.
8. Abnormal cytology on a cervical screening based on the American College of Obstetricians and Gynecologists (ACOG) guidelines and patient age. (CIN1 or HPV allowed to participate in the study, CIN2 excluded unless treated and cleared, CIN3 excluded).
9. History of malignancy within 5 years of the start of screening, except for treated basal cell carcinoma and squamous cell carcinoma of the skin.
10. Any thoughts of suicide in the last 12 months per self-report, or documented in the electronic medical record (EMR).
11. Hypersensitivity to the study drugs.
12. Planned surgical treatment of endometriosis or planned surgery in the abdominal-pelvic area within the duration of the trial.
13. Untreated abnormal prolactin or TSH
14. Any conditions that preclude pregnancy.
15. Patients with a known history of a low-trauma fracture or other risk factors for osteoporosis or bone loss.
16. Patients with cirrhosis or abnormal LFTs per self report or documented in the electronic medical record (EMR).

    * Exclusion criteria number 1,2, and 3 are not required to be met by individuals in the standard of care arm of the study. The study team will collect the information regarding whether the subject has used these drugs in the aforementioned time frame using the concomitant medication log and the individual will be allowed to participate in the study under the standard of care arm only.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 297 (Estimated)
Dates: Start 2024-03-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | Up to 15 months
  Live birth rate per participant is defined as live birth at ≥24 weeks of gestation.

SECONDARY OUTCOMES:
Fertilization rate | Up to 9 months
  Fertilization rate per participant is defined as the rate of [two pronuclei (2PN)]/[total number of oocytes injected or inseminated]
Number of embryos transferred | Up to 9 months
  Number of embryos transferred per participant
Implantation rate | Up to 9 months
  Implantation rate per participant is defined as the rate of (number of gestation sacs visible by Ultrasound) / (Number of Embryo Transfer),
Biochemical pregnancy rate | Up to 9 months
  Biochemical pregnancy rate per participant is defined as positive pregnancy test following embryo transfer
Clinical pregnancy rate | Up to 10 months
  Clinical pregnancy rate per participant is defined as ultrasound evidence of intrauterine gestational sac with fetal cardiac activity
Miscarriage rate | Up to 10 months
  Miscarriage rate among those who achieved pregnancy. Miscarriage is defined as pregnancy loss prior to viability scan and including those confirmed on ultrasound scan up to ≤23+6 weeks of gestation gestation.
Overall pregnancy complication rate | Up to 15 months
  Overall pregnancy complication rate among those who achieved pregnancy. Overall pregnancy complication including any of the following: preterm delivery, preeclampsia, incidence of abnormal placentation (placenta previa, accreta, increta, percreta, abruption), bleeding in pregnancy (antepartum or postpartum)
Gestation age at delivery | Up to 15 months
  Gestation age (weeks) at delivery per infant delivered
Infant birth weight | Up to 15 months
  Infant birth weight (gram) per infant delivered.

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Taylor, MD, Principal Investigator — Yale University; Heping Zhang, PhD, Study Director — Yale University; Nanette Santoro, MD, Study Director — University of Colorado, Denver; Emily Jungheim, MD, Study Director — Northwestern University; Steven Young, MD, PhD, Study Director — Duke University; Jim Segars, MD, Study Director — Johns Hopkins University
Locations (5):
- United States (5):
  - University of Colorado Department of Obstetrics & Gynecology, Aurora, Colorado
  - Yale School of Medicine Dept.of Ob/Gyn & Reproductive Sciences, New Haven, Connecticut
  - Northwestern University Department of Obstetrics and Gynecology, Chicago, Illinois
  - Johns Hopkins, Division of Reproductive Science and Women's Health Research, Baltimore, Maryland
  - Duke Fertility, Morrisville, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
The investigators have a plan to submit data and samples collected by the trial to NICHD DASH. The informed consent will include permission to bank these samples. The processes included initial data and documentation preparation (e.g., codebooks, protocols, informed consent for data sharing), data quality control, and submission.
Supporting Information: Study Protocol, SAP, ICF, CSR